CLINICAL TRIAL: NCT05686122
Title: Initial Testing of a Mobile App Pain Coping Intervention for Outpatient Oncology Settings
Brief Title: Initial Testing of a Mobile App Pain Coping Intervention for Outpatient Oncology Settings (PainPac)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00112397; 1R21CA273832 (NIH)
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer
Keywords: cancer; pain; coping; mHealth; symptom management
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PainPac (Experimental): 4 behavioral cancer pain intervention sessions delivered by mobile application. Patient-focused intervention. PainPac uses Social Cognitive Theory to promote behaviors to improve pain, self-efficacy for pain management, and pain-related quality of life indices. It also uses real-time data to personalize the intervention and messaging to participants. The app also has interactive components to improve coping skills engagement.
  Interventions: Behavioral: PainPac
- PCST-Video (No Intervention): 4 behavioral cancer pain intervention sessions delivered by videoconferencing by a pain therapist in the medical center to the patient in their natural environment (e.g., home). Sessions will be scheduled weekly for 45-60 min and mimic in person sessions. PCST-Video session content is matches the PainPac skills modules. PCST-Video participants will complete assessments at the same intervals as PainPac participants.

INTERVENTIONS:
Behavioral: PainPac — Patient-focused behavioral pain intervention delivered via mobile application.
  Arms: PainPac

SUMMARY:
PainPac is innovative in its potential to integrate with healthcare systems through electronic medical records (EMRs). PainPac leverages technology to increase patient access to interventions and uses real-time assessment to improve care. PainPac is positioned to rapidly provide improved care through combining biological data (e.g., EMRs, patient collected) with behavioral data to dramatically improve outcomes. PainPac could track beneficial outcomes related to clinical pain scores (e.g., patients with scores 4-8 benefit) and intervention implementation could be based on this; a more advanced possibility is use of geospatial tracking to predict space/time where pain is likely to impact functioning and push an intervention strategy - behavioral or pharmacological. PainPac is designed for future transmission of data to EMRs to inform providers of patient status. This work will provide data to bypass traditional efficacy trials and move quickly to a large effectiveness trial.

DETAILED DESCRIPTION:
The investigators will use a pilot RCT to examine PainPac feasibility, patient burden, engagement, acceptability, and initial pain-related outcomes, compared to a therapist led videoconference delivered behavioral pain intervention (PCST-Video) in colorectal cancer patients with pain. Investigators will use quantitative and qualitative data to optimize PainPac. Participants will complete assessments at pre-treatment (A1), post-treatment (A2; 4 weeks post-A1), and 1 month follow-up (A3; 1 month post-A2) (months 5-22). The pain management strategies are relevant and efficacious across cancer types. Due to the pilot nature of this work, investigators will enroll an opportunity sample of colorectal cancer patients.

PainPac is a patient-focused intervention developed using cognitive-behavioral theory and empirically supported strategies to enhance patients' ability to manage their pain. PainPac is a mobile app available to participants on a smartphone or tablet. PainPac uses Social Cognitive Theory to promote behaviors to improve pain, self-efficacy for pain management, and pain-related quality of life indices. It also uses real-time data to personalize the intervention and messaging to participants. PainPac contains 4 modules, each including a skill that has shown efficacy for reducing pain in patients with cancer. Patients are prompted to complete one module each week for 4 weeks. The app also has interactive components to improve coping skills engagement.

Participants randomized to PCST-Video will receive 4 behavioral cancer pain intervention sessions delivered by videoconferencing by a pain therapist in the medical center to the patient in their natural environment (e.g., home). Sessions will be scheduled weekly for 45-60 min and mimic in person sessions. PCST-Video session content is matches the PainPac skills modules described above. PCST-Video participants will complete assessments at the same intervals as PainPac participants.

Aim 1: Test whether PainPac is feasible (primary aim), low burden, engaging, and acceptable.

Aim 2: Examine the impact of PainPac on pain severity, pain interference, pain self-efficacy, and quality of life.

Aim 3: Gather quantitative and qualitative post-treatment data on patients' preferences, barriers, and facilitators regarding PainPac to update and optimize PainPac for a future large randomized clinical effectiveness trial.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-IV Colorectal Cancer diagnosis
* 18 years of age or older

Exclusion Criteria:

* Cognitive Impairment
* Brain Metastases
* Severe psychiatric condition (e.g., psychosis) that would contraindicate safe participation
* Participation in behavioral pain management in the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah A Kelleher, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two additional participants were consented but were not randomized and did not complete the baseline assessments.
Groups:
- PainPac: 4 behavioral cancer pain intervention sessions delivered by mobile application. Patient-focused intervention. PainPac uses Social Cognitive Theory to promote behaviors to improve pain, self-efficacy for pain management, and pain-related quality of life indices. It also uses real-time data to personalize the intervention and messaging to participants. The app also has interactive components to improve coping skills engagement.
  PainPac is a patient-focused behavioral pain intervention delivered via mobile application.
Period: Overall Study
Arm/Group | PainPac | PCST-Video
Started | 30 | 30
Completed | 28 | 30
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PainPac | PCST-Video | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 23 | 44
  >=65 years | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.10 (12.41) | 58.20 (10.46) | 58.15 (11.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 12 | 10 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 29 | 28 | 57
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 10 | 16
  White | 23 | 18 | 41
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Measured by Study Accrual
Description: Reaching target accrual (N=60) within 15 months.
Time Frame: Baseline
Population: Out of 82 patients who screened eligible for this study, 62 patients consented to participate. 60 of those patients completed the baseline assessment and were randomized.
Measure: Number; unit: participants
Groups:
- Total Consented Participants: Out of 82 patients who screened eligible for this study, 62 patients consented to participate. 60 of those patients completed the baseline assessment and were randomized.
Arm/Group | Total Consented Participants
Number analyzed (Participants) | 82
participants | 62

2. Primary Outcome: Feasibility as Measured by Attrition (Number of Participants Who Did Not Complete the 1-month Visit)
Time Frame: 1-month follow-up (9-12 weeks post-baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | PainPac | PCST-Video
Number analyzed (Participants) | 30 | 30
Participants | 2 | 1

3. Primary Outcome: Feasibility as Measured by the Number of Participants Who Completed Study Baseline Assessments
Description: Protocol adherence indicated by calculating the degree to which participants are willing/able to complete the study baseline assessment.
Time Frame: Baseline
Population: The number analyzed for this outcome includes the two participants who consented but did not complete the baseline assessments and were not randomized. Since the baseline assessment occurs before randomization, the study groups are combined for this measure.
Measure: Count of Participants; unit: Participants
Groups:
- Total Consented Participants: All participants who consented to the study, regardless of baseline completion
Arm/Group | Total Consented Participants
Number analyzed (Participants) | 62
Participants | 60

4. Primary Outcome: Feasibility as Measured by the Number of Participants Who Completed Post-study Sessions Assessments
Description: Protocol adherence indicated by calculating the degree to which participants are willing/able to complete the post-study sessions assessment.
Time Frame: Post-treatment assessment (5-8 weeks post-baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | PainPac | PCST-Video
Number analyzed (Participants) | 30 | 30
Participants | 28 | 27

5. Primary Outcome: Feasibility as Measured by the Number of Participants Who Completed Study 1-month Follow up Assessments Completed
Description: Protocol adherence indicated by calculating the degree to which participants are willing/able to complete the 1-month follow up assessment.
Time Frame: 1-month follow-up (9-12 weeks post-baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | PainPac | PCST-Video
Number analyzed (Participants) | 30 | 30
Participants | 28 | 29

6. Primary Outcome: Feasibility of PainPac, as Measured by the Total # of Participants Who Completed All Four Sessions
Description: Includes protocol adherence indicated by calculating the degree to which participants are willing/able to complete the 4 PainPac skills modules or 4 PCST-Video sessions.
Time Frame: 5-8 weeks post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | PainPac | PCST-Video
Number analyzed (Participants) | 30 | 30
Participants | 27 | 24

7. Secondary Outcome: Acceptability as Measured by the Client Satisfaction Questionnaire.
Description: 10-item Client Satisfaction Questionnaire (CSQ). This questionnaire contains 10 items rated from 1=low acceptability to 4=high acceptability; scores are created by utilizing the Likert Scale to average Client Satisfaction Questionnaire answers resulting in a score range from 1-4. The participant will complete this acceptability questionnaire as part of the post-session follow up assessment. A higher score indicates a higher satisfaction, with 32 indicating 100% satisfaction and 8 indicating 0% satisfaction.
Time Frame: Post-treatment assessment (5-8 weeks post-baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PainPac | PCST-Video
Number analyzed (Participants) | 30 | 30
units on a scale | 28.11 (3.74) | 28.93 (3.57)

8. Secondary Outcome: Acceptability as Measured by Atkinson's Tool of mHealth Innovations.
Description: Atkinson's tool will also be used to assess perceived attributes of mHealth innovations. Tool has 30 items about mHealth, participant indicates their level of agreement or disagreement on a 6-point Likert scale: l=strongly disagree, 2=disagree, 3=somewhat disagree, 4=somewhat agree. 5=agree, and 6=strongly agree. Scores range from 1-6 with higher scores indicating a more positive assessment of PainPac.
Time Frame: Post-treatment assessment (5-8 weeks post-baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- PainPac: Participants who completed sessions via mobile application
Arm/Group | PainPac
Number analyzed (Participants) | 30
units on a scale | 4.82 (.52)

9. Secondary Outcome: Computer Self-Efficacy
Description: Post-Intervention, 10 items on a 10 point scale from 0=not at all confident to 10=completely confident. Total score ranges from 0-100. Patients are asked 10 items regarding their confidence in ability to use technology (computer and smartphone app). Higher scores indicate greater computer self-efficacy.
Time Frame: Post-treatment assessment (5-8 weeks post-baseline)
Population: Computer Self-Efficacy was a PainPac-specific measure of self-efficacy, and thus only PainPac participants completed this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PainPac
Number analyzed (Participants) | 28
score on a scale | 83.71 (19.82)

10. Secondary Outcome: Change in Pain Severity as Assessed With the Brief Pain Inventory (BPI)
Description: Pain will be assessed with the Brief Pain Inventory (BPI). Patients will rate their "worst", "least", "average", and "now" pain from 0=no pain to 10=worst pain imaginable. An average of the responses to these items is used to create a single pain severity score.
Time Frame: Baseline, Post-Assessment (5-8 weeks post-baseline), 1 month follow-up (9-12 weeks post-baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PainPac | PCST-Video
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline (A1) | 3.73 (1.91) | 4.55 (2.32)
  Post-Assessment (A2) | 3.88 (1.88) | 3.96 (2.19)
  1 month follow-up (A3) | 3.51 (2.49) | 3.37 (2.10)

11. Secondary Outcome: Pain Interference as Assessed With the Brief Pain Inventory (BPI) - Pain Interference Scale
Description: Pain interference will be assessed with the Brief Pain Inventory (BPI) - Pain Interference Scale. Patients will rate how much pain interfered with a variety of activities and mood states over the last 7 days from 0=does not interfere to 10=completely interferes. An average of the responses to these items is used to create a single pain severity score ranging from 0-10.
Time Frame: Baseline, Post-Assessment (5-8 weeks post-baseline), 1 month follow-up (9-12 weeks post-baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PainPac | PCST-Video
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline (A1) | 3.34 (2.07) | 4.08 (2.55)
  Post-Assessment (A2) | 3.05 (1.69) | 3.21 (2.19)
  1-month follow-up (A3) | 2.78 (2.12) | 2.77 (2.07)

12. Secondary Outcome: Change in Pain Self-Efficacy for Pain Management
Description: 5-item self-efficacy subscale of the Chronic Pain Self-Efficacy Scale. Items ask about patients' certainty about pain control, pain during activities, and reducing pain without extra medication using a 10=very uncertain to 100=very certain scale and averaged. Total score ranges from 10-100. Higher scores correspond to higher self-efficacy for pain management.
Time Frame: Baseline, Post-Assessment (5-8 weeks post-baseline), 1 month follow-up (9-12 weeks post-baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PainPac | PCST-Video
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline (A1) | 53.72 (23.69) | 59.70 (23.08)
  Post-Assessment (A2) | 63.79 (16.72) | 67.92 (21.32)
  1-month follow-up (A3) | 67.00 (20.40) | 65.52 (22.61)

13. Secondary Outcome: Burden as Measured by # of Sessions Completed
Time Frame: 3-8 weeks post-baseline
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | PainPac | PCST-Video
Number analyzed (Participants) | 30 | 30
sessions | 3.77 (.82) | 3.37 (1.33)

14. Secondary Outcome: Burden as Measured by # of Days From the Baseline Assessment to Completion of Session 1 (Days to Start Intervention)
Time Frame: 0-2 weeks post-baseline
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PainPac | PCST-Video
Number analyzed (Participants) | 30 | 30
days | 1.32 (2.28) | 12.25 (10.92)

15. Secondary Outcome: Burden as Measured by # of Days to Complete All Modules/Sessions (Days to Complete Intervention)
Time Frame: 3-8 weeks from Session 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PainPac | PCST-Video
Number analyzed (Participants) | 30 | 30
days | 23.57 (5.31) | 27.63 (6.70)

16. Secondary Outcome: Engagement in Study
Description: Engagement is defined as the number of times/week participants log into PainPac and practice the skills. Engagement will be assessed based on app data and patient self-report. Patient Engagement will be assessed by electronic app data (e.g., PainPac weekly log-ins) and patient self-report defined as the number of times per week they practice the coping skills. >3 times/week will serve as the benchmark; if participants log into PainPac and/or practice the coping skills <3 times/week, PainPac will not be considered engaging.
Time Frame: 5-8 weeks post-baseline
Population: Patients in the PCST-Video arm did not log into a mobile app so were not analyzed for the number of weekly log ins.
Measure: Mean (Standard Deviation); unit: Times per week
Groups:
- PCST-Video: Participants who completed sessions via videoconferencing
Arm/Group | PainPac | PCST-Video
Number analyzed (Participants) | 30 | 30
Times per week
  Weekly Log-Ins: number analyzed (Participants) | 30 | 0
  Weekly Log-Ins | 9.22 (4.20) |
  Weekly Skills Practice | 5.21 (1.91) | 5.52 (1.63)

17. Secondary Outcome: Change in Quality of Life
Description: This measure assesses healthy days in the last month.
Time Frame: Baseline, Post-Assessment (5-8 weeks post-baseline), 1 month follow-up (9-12 weeks post-baseline)
Measure: Mean (Standard Deviation); unit: healthy days in the past month
Arm/Group | PainPac | PCST-Video
Number analyzed (Participants) | 30 | 30
healthy days in the past month
  Baseline (A1) | 6.66 (7.18) | 9.60 (9.50)
  Post-assessment (A2) | 7.39 (7.49) | 8.63 (8.85)
  1-month follow-up (A3) | 9.50 (9.28) | 14.93 (15.27)

18. Secondary Outcome: Change in PROMIS - Emotional Distress (Depression) Short Form
Description: Post-intervention and 1-month follow up, 8 items on a 5 point scale from 1=never, 2=rarely, 3=sometimes, 4=often, 5=always. Patients are asked 8-items regarding "in the past 7 days I felt..." to assess their emotional distress levels. The total score ranges from 37.1-81.1, with higher scores indicate higher distress.
Time Frame: Baseline, Post-Assessment (5-8 weeks post-baseline), 1 month follow-up (9-12 weeks post-baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PainPac | PCST-Video
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline (A1) | 51.19 (7.13) | 50.16 (8.65)
  Post-Assessment (A2) | 50.52 (7.11) | 47.43 (8.98)
  1-month follow-up (A3) | 49.20 (8.34) | 48.24 (10.23)

ADVERSE EVENTS:
Time Frame: Approximately 11 weeks
Arm/Group | PainPac | PCST-Video
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-03): https://cdn.clinicaltrials.gov/large-docs/22/NCT05686122/Prot_SAP_001.pdf
  • Informed Consent Form (2024-03-14): https://cdn.clinicaltrials.gov/large-docs/22/NCT05686122/ICF_002.pdf